CLINICAL TRIAL: NCT04907721
Title: Development and Evaluation of a Glucagon Sensitivity Test in Individuals With and Without Hepatic Steatosis
Acronym: GLUSENTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Bispebjerg Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nicolai Jacob Wewer Albrechtsen, Associate Professor, MD, PhD, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GLUSENTIC
Record Dates: First submitted 2021-05-17; First posted 2021-06-01 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Glucagon Resistance; Type 1 Diabetes; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 1; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measuring glucagon sensitivity in humans (Experimental): Participants will be subjected to two experimental days.
  Interventions: Diagnostic Test: Glucagon Sensitivity test consisting of an amino acid tolerance test and a bolus infusion of glucagon

INTERVENTIONS:
Diagnostic Test: Glucagon Sensitivity test consisting of an amino acid tolerance test and a bolus infusion of glucagon — The test consists of two experimental study days:
  Day 1: intravenous bolus-injection of glucagon (0.2 mg at time 0 minutes) evaluating the effect of exogenous glucagon on amino acid disappearance. Blood samples will be obtained from time -10 to 120 minutes.
  Day 2: 45-minute intravenous infusion of mixed amino acids (331 mg/min/kg body weight from time 0-45 minutes) to evaluate the effect of endogenous glucagon on amino acid metabolism. Blood samples will be obtained from time -10 to 180 minutes.
  All participants will be subjected to a magnetic resonance imaging scan to assess whole-liver steatosis, and a bioelectrical impedance analysis to assess body composition.
  Following study inclusion and the magnetic resonance imaging scan, participants will be stratified into groups based on hepatic steatosis. Individuals with <5.6 % hepatic steatosis will be classified as controls and individuals with ≥5.6 % hepatic steatosis will be classified as MASLD.

SUMMARY:
Glucagon is secreted from pancreatic alpha-cells in response to protein-rich meals and during hypoglycemia. A physiological feedback system exists between the liver and the pancreatic alpha cells termed the liver-alpha cell axis and signifies the role between amino acid-stimulated glucagon secretion and glucagon-stimulated amino acid metabolism.

Individuals with non-alcoholic fatty liver disease have increased levels of glucagon (hyperglucagonemia) and amino acids (hyperaminoacidemia), which suggests that hepatic steatosis may uncouple glucagon's effect on amino acid metabolism (i.e. reduced glucagon sensitivity). Since hyperglucagonemia contributes to diabetes progression - due to its potentiating effects on hepatic glucose production - hepatic steatosis may create a diabetogenic circle. This study aims to develop and evaluate a test for measuring glucagon sensitivity in humans.

The investigators (Associate Prof. Nicolai J Wewer Albrechtsen and Prof. Jørgen Rungby) will investigate whether amino acid metabolism is attenuated in individuals with hepatic steatosis (assessed by magnetic resonance imaging) due to impaired hepatic glucagon sensitivity and if glucagon's effect on hepatic glucose production is intact compared to individuals without hepatic steatosis suggestive of biased signaling.

DETAILED DESCRIPTION:
Amino acids administered orally or intravenously stimulate glucagon secretion from the pancreas and in turn, glucagon is a powerful stimulus for hepatic amino acid turnover through transcriptional (long-term) and non- transcriptional (acute) mechanisms. Several groups including the investigators have linked glucagon secretion to hepatic amino acid metabolism suggesting a mutual feedback cycle, termed the liver-alpha cell axis. A disruption of this axis, which has been shown both pharmacologically using glucagon receptor antagonists and genetically in glucagon receptor knockout mouse models, leads to increased glucagon (hyperglucagonemia) and amino acid (hyperaminoacidemia) concentrations. This phenotype is also evident in subjects with biopsy-verified metabolic dysfunction-associated steatotic liver disease (MASLD) independent of type 2 diabetes suggesting reduced hepatic glucagon sensitivity in the presence of hepatic steatosis. Glucagon increases amino acid catabolism by potentiating ureagenesis, a pathway exclusive to the liver, and hepatic accumulation of triglycerides may reduce glucagon's ability to augment amino acid turnover. Some amino acids are more potent in stimulating glucagon secretion (glucagonotropic amino acids), including alanine, and the glucagon-alanine index is currently used as a surrogate marker for the hepatic actions of glucagon on ureagenesis. The fate of amino acid turnover depends on both glucagon and insulin dynamics by stimulating amino acid catabolism and synthesis, respectively. Studying the effects of glucagon in individuals with type 1 diabetes will allow one to differentiate between the combined effects of glucagon and insulin compared to the effects of glucagon alone.

This study aims to explore hepatic glucagon sensitivity towards amino acid metabolism in individuals with and without hepatic steatosis (based on magnetic resonance imaging (MRI)).

The investigators hypothesize that the effect of endogenous and exogenous glucagon on plasma amino acid levels are impaired in individuals with MASLD (based on hepatic steatosis measured by MRI) compared to controls.

The nomenclature for MASLD has recently been updated from non-alcoholic fatty liver disease (NAFLD) (https://pubmed.ncbi.nlm.nih.gov/37363821/).

ELIGIBILITY:
Group 1 (lean controls)

Inclusion Criteria:

* BMI = 18.6-25 kg/m2
* Male or female
* 25-65 years of age

Exclusion Criteria:

* Diabetes (ADA criteria)
* Significant alcohol/drug abuse as per investigators judgement
* Amino acid-related diseases such as phenylketonuria
* Kidney disease
* Cardiac problems
* Cancer within the past 1 year
* Severe claustrophobia
* Pacemaker or other non-MR-compatible devices
* Pregnancy or breastfeeding.
* Fib4 score > 3.25.
* Any medicine, acute illness (within the last two weeks) or other circumstances that in the opinion of the investigator might endanger the participants' safety or compliance with the protocol

Group 2 (overweight and obese individuals)

Inclusion Criteria:

* BMI = 25-40 kg/m2
* Male or female
* 25-65 years of age

Exclusion Criteria:

* Diabetes (ADA criteria)
* Significant alcohol/drug abuse as per investigators judgement
* Amino acid-related diseases such as phenylketonuria
* Kidney disease
* Cardiac problems
* Cancer within the past 1 year
* Severe claustrophobia
* Pacemaker or other non-MR-compatible devices
* Pregnancy or breastfeeding
* Abdominal diameter >70 cm
* Fib4 score > 3.25.
* Any medicine, acute illness (within the last two weeks) or other circumstances that in the opinion of the investigator might endanger the participants' safety or compliance with the protocol

Group 3 (individuals with type 1 diabetes)

Inclusion Criteria:

* BMI = 18.6-40 kg/m2
* Male or female
* C-peptide negative
* Insulin pump user
* 25-65 years of age

Exclusion Criteria:

* Type 2 diabetes
* Closed loop user
* Microalbuminuria (30-300 mg/g)
* Significant alcohol/drug abuse as per investigators judgement
* Amino acid-related diseases such as phenylketonuria
* Kidney disease
* Cardiac problems
* Cancer within the past 1 year
* Severe claustrophobia
* Pacemaker or other non-MR-compatible devices
* Pregnancy or breastfeeding
* Abdominal diameter >70 cm
* Fib4 score > 3.25.
* Any medicine, acute illness (within the last two weeks) or other circumstances that in the opinion of the investigator might endanger the participants' safety or compliance with the protocol

Following inclusion and study completion, our two groups of lean individuals (n=20) and overweight and obese individuals (n=30) will be stratified into two groups based on liver fat content assessed by the magnetic resonance imaging scan. Individuals with <5.6% hepatic steatosis will be allocated to the control group and individuals with ≥5.6% hepatic steatosis to the MASLD group.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2023-10-21 (Actual)

PRIMARY OUTCOMES:
Differences in the calculated GLUSENTIC index between individuals with or without MASLD without diabetes | Time from the first blood sample (at time -10 minutes, following an overnight fast) until the amino acid infusion stops (45 minutes)
  This index is conceptually be based on the Matsuda/composite index, and will factor in fasting and amino acid-stimulated levels of glucagon and total amino acids using the following formula: 100/(SQRT(Fasting plasma amino acids levels (mean at time -10 and 0 minutes) * Fasting plasma glucagon levels (mean at time -10 and 0 minutes) * Amino acid-stimulated amino acid levels (mean at time 40 and 45 minutes) * Amino acid-stimulated glucagon levels (mean at time 40 and 45 minutes)).

SECONDARY OUTCOMES:
Simple linear regression between hepatic steatosis (%) and the GLUSENTIC index | Time from the first blood sample (at time -10 minutes, following an overnight fast) until the amino acid infusion stops (45 minutes)
  Measurements of hepatic steatosis will be assessed by magnetic resonance imaging. Data from controls and MASLD without diabetes will be included.
ROC curve analysis to evaluate cut-off value for GLUSENTIC index | Time from the first blood sample (at time -10 minutes, following an overnight fast) until the amino acid infusion stops (45 minutes)
  Controls and MASLD groups will be included.
Differences in the glucagon-alanine index | The index will be measured on samples collected after an overnight fast (12 hours)
  The glucagon-alanine index will be measured as previously described: https://pubmed.ncbi.nlm.nih.gov/29305624/. Measurements of hepatic steatosis will be assessed by magnetic resonance imaging. Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Differences in plasma levels of amino acids during the amino acid tolerance test (determined by baseline corrected AUC) | Time from the start of infusion (0 minutes) until time 60 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Glucagon's ability (exogenous glucagon) to increase amino acid disappearance (determined by baseline corrected AUC or delta) for total amino acid levels and the individual amino acids. | Time from the glucagon injection (time 0 minutes) until time 20 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Differences in plasma levels of total amino acids and alanine following an overnight fast. | Measured on samples collected after an overnight fast (12 hours)
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Baseline corrected AUC for glucagon after a bolus injection of glucagon. | Time from the glucagon injection (time 0 minutes) until time 120 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Baseline corrected AUC for glucagon during and after the amino acid tolerance test. | Time from the amino acid infusion starts (time 0 minutes) until time 180 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made. For insulin and C-peptide measurements, only individuals without diabetes will be compared.
Differences in plasma levels of glucagon following an overnight fast. | Measured on samples collected after an overnight fast (12 hours)
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Baseline corrected AUC for glucose after a bolus injection of glucagon. | Time from the glucagon injection (time 0 minutes) until time 120 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Baseline corrected AUC for insulin after a bolus injection of glucagon. | Time from the glucagon injection (time 0 minutes) until time 120 minutes.
  Comparisons between controls and MASLD will be made.
Baseline corrected AUC for C-peptide after a bolus injection of glucagon. | Time from the glucagon injection (time 0 minutes) until time 120 minutes.
  Comparisons between controls and MASLD will be made.
Baseline corrected AUC for urea after a bolus injection of glucagon. | Time from the glucagon injection (time 0 minutes) until time 120 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Baseline corrected AUC for triglycerides after a bolus injection of glucagon. | Time from the glucagon injection (time 0 minutes) until time 120 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Baseline corrected AUC for glucose during and after the amino acid tolerance test. | Time from the amino acid infusion starts (time 0 minutes) until time 180 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Baseline corrected AUC for insulin during and after the amino acid tolerance test. | Time from the amino acid infusion starts (time 0 minutes) until time 180 minutes.
  Comparisons between controls and MASLD will be made.
Baseline corrected AUC for C-peptide during and after the amino acid tolerance test. | Time from the amino acid infusion starts (time 0 minutes) until time 180 minutes.
  Comparisons between controls and MASLD and will be made.
Baseline corrected AUC for urea during and after the amino acid tolerance test. | Time from the amino acid infusion starts (time 0 minutes) until time 180 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Baseline corrected AUC for triglycerides during and after the amino acid tolerance test. | Time from the amino acid infusion starts (time 0 minutes) until time 180 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Differences in the formula (plasma urea/plasma amino acids) after the amino acid tolerance test. | Time from the amino acid infusion stops (time 45 minutes) until time 180 minutes.
  Comparisons between controls, MASLD and individuals with type 1 diabetes will be made.
Differences in total and individual amino acids between individuals with overweight or obesity without hepatic steatosis who have been BMI-matched to individuals with hepatic steatosis. | Time 0-120 minutes on the day of the glucagon injection and time 0-180 minutes on the day of the amino acid tolerance test.
  Baseline subtracted AUCs will be made and individuals with or without MASLD, who are matched on BMI in a 1:2 ratio will be compared.
Differences in glucagon between individuals with overweight or obesity without hepatic steatosis who have been BMI-matched to individuals with hepatic steatosis. | Time time 0-180 minutes on the day of the amino acid tolerance test.
  Baseline subtracted AUCs will be made and individuals with or without MASLD, who are matched on BMI in a 1:2 ratio will be compared.
Simple linear regression between the variables, pancreatic steatosis and amino acid stimulated glucagon or insulin levels in individuals without diabetes. | Pancreatic steatosis and time point 30 minutes on the day of the amino acid tolerance test will be used.
  Data from controls and MASLD will be included.

OTHER OUTCOMES:
Differences in FGF-21 | From time -10 to 120 minutes on the day of the glucagon bolus infusion and from time -10 to 180 minuteson the day of the amino acid infusion.
  Comparisons between controls, individuals with hepatic steatosis and individuals with type 1 diabetes will be made.
Differences in GLP-1 | From time -10 to 120 minutes on the day of the glucagon bolus infusion and from time -10 to 180 minutes on the day of the amino acid infusion.
  Comparisons between controls, individuals with hepatic steatosis and individuals with type 1 diabetes will be made.
Differences in GIP | From time -10 to 120 minutes on the day of the glucagon bolus infusion and from time -10 to 180 minutes on the day of the amino acid infusion.
  Comparisons between controls, individuals with hepatic steatosis and individuals with type 1 diabetes will be made.
Differences in GDF-15 | From time -10 to 120 minutes on the day of the glucagon bolus infusion and from time -10 to 180 minutes on the day of the amino acid infusion.
  Comparisons between controls, individuals with hepatic steatosis and individuals with type 1 diabetes will be made.
Differences in focused genotyping (PNPLA3; MBOAT7; GCKR; TNF; TM6SF2). | From time -10 to 120 minutes on the day of the glucagon bolus infusion and from time -10 to 180 minutes on the day of the amino acid infusion.
  Comparisons between controls, individuals with hepatic steatosis and individuals with type 1 diabetes will be made.
Differences in follistatin | From time -10 to 120 minutes on the day of the glucagon bolus infusion and from time -10 to 180 minuteson the day of the amino acid infusion.
  Comparisons between controls, individuals with hepatic steatosis and individuals with type 1 diabetes will be made.
Differences in fetuin-B | From time -10 to 120 minutes on the day of the glucagon bolus infusion and from time -10 to 180 minuteson the day of the amino acid infusion.
  Comparisons between controls, individuals with hepatic steatosis and individuals with type 1 diabetes will be made.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
We have not decided to share IPD as this also would require approval from the ethical and data approval comitee.

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT04907721/SAP_002.pdf